CLINICAL TRIAL: NCT00104377
Title: A Multicenter, Single-Blind, Placebo-Controlled, Phase 2 Study to Evaluate the Induction of Immunogenicity With Different Doses of Grass MATA in Subjects Allergic to Grass and Rye Pollen
Brief Title: Induction of Immunogenicity With Different Doses of Grass MATA in Subjects Allergic to Grass and Rye Pollen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GrassMATAMPL201
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2009-09

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Allergoid; Specific Immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: Grass MATA MPL

SUMMARY:
Grass MATA (modified pollen allergen tyrosine adsorbate) has been developed to provide pre-seasonal specific immunotherapy for patients with hypersensitivity to grass and rye pollen. Different doses of Grass MATA will be administered and immunological changes following this treatment will be assessed.

DETAILED DESCRIPTION:
Grass MATA MPL has been developed to provide pre-seasonal specific immunotherapy for patients with proven type I hypersensitivity to cross reacting grass pollens.

The grass pollen extract is modified with glutaraldehyde to produce the active ingredient, an allergoid. This modification reduces the reactivity of the extract with IgE antibody, thus reducing the risk of side effects. However, a simultaneous reduction in other important immunological properties, such as IgG and T cell reactivities, is not seen.

MPL (Monophosphoryl Lipid A), a purified, detoxified glycolipid derived from the cell wall of Salmonella minnesota, is included in the product formulation as an adjuvant to increase the immunogenic effect of the product and to enhance the switch from an allergen-specific TH2 to a TH1-like T cell profile.

The purpose of this study is to assess specific immunological changes (IgG, IgG1, IgG4 and IgE) in allergic subjects following 2 subcutaneous injections of different doses of study medication (Grass MATA or placebo) administered 3 weeks apart. The immunological changes will be used to assess the performance of the R7 IgG reactivity assay over a range of clinically efficacious doses.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential may enter the study if they have a negative urine pregnancy test and they have been practicing adequate contraception for 3 months prior to the study and continue to do so during the study
* History of at least 1 season of moderate to severe seasonal rhinoconjunctivitis without bronchial asthma due to an IgE mediated allergy to pollen from grasses and rye
* Positive skin prick test to grass pollen and to rye pollen allergen extract
* Positive skin prick test to positive histamine control
* Negative skin prick test to negative control
* Specific IgE for grass and rye as documented by a RAST or equivalent test
* Moderate/severe allergy symptoms in the past spring season
* Spirometry at Screening demonstrates FEV1 >= 80% predicted and FEV1/FVC >= 70%.

Exclusion Criteria:

* History or presence of acute or subacute atopic dermatitis, chronic dermatitis, urticaria factitia, or urticaria due to physical/chemical influence or any other skin conditions which might interfere with the interpretation of skin prick test results
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the screening skin prick tests; both forearms must be available for testing
* History of bronchial asthma, chronic obstructive pulmonary disease (COPD), or other chronic condition of the lower respiratory tract
* History or presence of diabetes (insulin dependent and non-dependent), cancer or any clinically significant cardiac, metabolic, renal, hepatic, gastrointestinal, dermatologic, venereal, hematologic, neurologic or psychiatric diseases or disorders
* Any clinically significant abnormal laboratory value at Visit 1
* Clinically relevant sensitivity to any common perennial allergen: house dust mites, molds, or epithelia (cat, dog, and horse). Subjects may be enrolled in the study if they test positive (skin prick test or RAST), but have no current or historical symptoms to perennial allergens.
* Clinically relevant sensitivity to any common springtime flowering plant: Birch, Oak, Sycamore, Beech, Ash and Poplar. Subjects may be enrolled in the study if they test positive (skin prick test or RAST), but have no current or historical symptoms to these springtime allergens.
* History of auto-immune diseases or rheumatoid diseases
* Subject not allowed to receive adrenalin
* Subject has disorder of tyrosine metabolism (i.e., alcaptonuria, tyrosinemia)
* Subject with diseases interfering with the immune response and have received medication, which could influence the results of this study
* Subject has acute or chronic infection
* History of anaphylaxis, including anaphylactic food allergy, insect venom anaphylaxis, exercise or drug induced anaphylaxis
* History of angioedema
* History of hypersensitivity to the excipients of the study medication
* History of immunotherapy with grass allergen extracts
* Current therapy with ß-blockers
* Currently receiving anti-allergy medication or other medications with an antihistaminic activity
* Subject has a positive drugs of abuse screen at Visit 1
* Subject participated in a clinical trial with an investigational medication within the last 3 months
* Subject cannot communicate reliably with the Investigator or is not likely to cooperate with the requirements of the study
* Subject is pregnant or lactating
* Use of prohibited medications or inadequate washout periods prior to screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
To assess specific immunological changes (IgG, IgG1, IgG4, IgE) in grass and rye allergic subjects following 2 subcutaneous injections of study medication (different doses of Grass MATA or placebo) administered 3 weeks apart.

SECONDARY OUTCOMES:
adverse events
clinical laboratory evaluations
vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Paul H. Ratner, MD, Principal Investigator — Sylvana Research Associates
Locations (11):
- United States (11):
  - College Park Family Care Center Multi-Specialty Clinical Research, Overland Park, Kansas
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Midwest Clinical research, LLC, St Louis, Missouri
  - Allergy, Asthma, and Immunology Assoc. PC, Lincoln, Nebraska
  - Asthma, Sinus, and Allergy Centers, LLC, Tinton Falls, New Jersey
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - Sylvana Research Associates, San Antonio, Texas